CLINICAL TRIAL: NCT04966390
Title: A Prospective,Multicenter,Non-interventional Real-world Study for Standardized Clinical Application of Antibacterial/Anitifungal Drugs
Brief Title: Standardized Clinical Application of Antibacterial/Anitifungal Drugs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, An Youzhong, Director of intensive care unit, Peking University People's Hospital
Other Study IDs: ANTI
Record Dates: First submitted 2021-07-14; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Antibiotics
Keywords: antibacterial/anitifungal drugs; real world study; standardized treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this real world study is to observe the clinical status for standardized using of antibacterial/anitifungal drugs in patients with infection,and to evaluate the efficacy and safety of anti-infection therapy.

DETAILED DESCRIPTION:
This study is a prospective,multicenter,non-interventional real-world study.The purpose of this study is to observe the clinical status of infection patients under standardized application of antibacterial/anitifungal drugs,and to evaluate the efficacy and safety of anti-infection treatment.

This study plans to enroll 5000 hospitalized patients (≥ 18 years old with infectious disease),who take antibacterial/anitifungal drugs for more than 3 days. Patients mainly come from ICU,Respiratory Department and Hematology Department.

The clinical data collection is divided into five parts,including Baseline,3rd and 7th day after the first dosing of antibacterial/anitifungal drugs,End of antibacterial/anitifungal drugs treatment (EOT),14th day after EOT. The collected clinical data cover general characteristics,condition assessment and severity evaluation,pathogenic diagnosis,the use of antibacterial/antifungal drugs,antibacterial/antifungal drugs-related adverse events,et al.

After completing the collection of case data, the proportion analysis, efficacy evaluation and safety evaluation for the standardized application of antibacterial/antifungal drugs will be carried out.

ELIGIBILITY:
Inclusion Criteria:

- Hospitalized patients (≥ 18 years old)

-≥ 3 days receiving antibacterial/antifungal drugs therapy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research plans to enroll 5000 hospitalized patients (≥ 18 years old with infectious disease), who use antibacterial/antifungal drugs for more than 3 days. Patients mainly come from ICU, respiratory department and hematology department.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-07-20 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of standardized using of antibacterial/antifungal drugs | approximately 6 months after completion of data collection
  the proportion of cases who receive standardized antibacterial/antifungal drugs therapy
Clinical efficacy rate | approximately 6 months after completion of data collection
  the clinical efficacy evaluation of antibacterial/antifungal drugs therapy

SECONDARY OUTCOMES:
Microbiological efficacy rate | approximately 6 months after completion of data collection
  the microbiological efficacy evaluation of antibacterial/antifungal drugs therapy
Overall efficacy rate | approximately 6 months after completion of data collection
  the overall efficacy evaluation of antibacterial/antifungal drugs therapy based on clinical and microbiological efficacy outcome
All-cause mortality | approximately 6 months after completion of data collection
  the evaluation of all-cause mortality
Antibacterial/antifungal drugs-Related Adverse Events | approximately 6 months after completion of data collection
  only evaluate of the adverse events related to antibacterial/antifungal drugs

CONTACTS AND LOCATIONS:
Overall Officials: Youzhong An, Principal Investigator — Peking University People 's Hospital